CLINICAL TRIAL: NCT01502605
Title: Phase I Study of Orally Administered Aminolevulinic Acid for Resection of Malignant Astrocytomas
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: PI leaving institution
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: J1140
Record Dates: First submitted 2011-12-29; First posted 2011-12-30 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Astrocytoma; Glioma
Keywords: 5-ALA; Aminolevulinic Acid; Craniotomy; Brain Tumor; Surgical Resection; Neurosurgery
MeSH Terms: conditions — Astrocytoma; Glioma; Brain Neoplasms | interventions — Aminolevulinic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 5-ALA (Experimental): This arm will receive the investigational agent, 5-ALA.
  Interventions: Drug: 5-Aminolevulinic Acid

INTERVENTIONS:
Drug: 5-Aminolevulinic Acid — A one time, single-dose administration of ALA is planned 4 hours pre-operatively the day of surgery. ALA will be mixed in the minimum volume of sterile water or juice immediately before use and given as a single oral bolus. Once ALA has been administered, patients will be kept in subdued lighting away from sunlight.

SUMMARY:
This research is being done to study the safety and utility of 5-aminolevulinic acid (5-ALA) (also known as Gliolan) for identifying brain tumor tissue during surgery. The goal of this study is to determine if 5-ALA can differentiate between tumor and normal brain tissue.

Sometimes, during brain surgery, the removal of tumor tissue can be difficult because the tumor can look like normal brain tissue. Studies in other countries have shown that in some brain tumors, 5-ALA can make the tumors appear brighter under ultraviolet light. This may make it easier for doctors to remove as much tumor as safely as possible from your brain.

This study also hopes to see if 5-ALA can find different cell populations within the tumor that is removed and allow the researchers to better understand brain tumors.

The purpose of this study is to:

* Find out how well 5-ALA can separate normal brain tissue from tumor tissues AND to see how well 5-ALA can find different cell populations within brain tumors
* Identify the amount of 5-ALA that should be taken before surgery to make the tumors glow under ultraviolet light
* Make sure the 5-ALA identifies tumor and not normal brain
* Make sure 5-ALA does not cause any side effects

ELIGIBILITY:
Inclusion Criteria:

* Patients must have clinically documented primary brain tumor for which resection is clinically indicated. Radiographic findings should be consistent with high grade glioma. Intraoperative frozen section should either be: anaplastic astrocytoma (WHO Grade III astrocytoma) or glioblastoma (WHO Grade IV astrocytoma).
* Patients must be aged greater than 18 years old
* Karnofsky Performance Score > 70 (Appendix)
* Patients must have normal organ and marrow function as defined below:

  * Leukocytes > 3,000 /uL
  * Absolute neutrophil count > 1,500/uL
  * Platelets > 100,000/uL
  * Total bilirubin within normal institutional limits
  * AST/ALT within normal institutional limits
  * Creatinine within normal institutional limits

Exclusion Criteria:

* Prior craniotomy for resection, deep seated tumors in thalamus and brain stem.
* History of allergic reactions to compounds of similar chemical composition to ALA.
* Personal or family history of porphyrias
* Personal history of hepatitis or other liver diseases.
* Pregnant women are excluded from this study because ALA is of unknown teratogenic effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with ALA, breastfeeding should be discontinued prior to treatment with ALA.
* Inability to undergo magnetic resonance imaging (i.e. those patients with AICD/pacemakers).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-09; Primary Completion 2015-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
serious adverse event (SAE) Rate | 2 weeks from dosing
  It will be considered as a serious adverse event with possible, probable, and definitely attribution to 5-ALA (SAE, detailed in section 8) if (within 2 weeks of dosing):
  Grade 1 or 2 LFT abnormalities not resolving within 2 weeks A single documented Grade 3 or 4 LFT abnormalities A Grade 3 or 4 skin photosensitivity

SECONDARY OUTCOMES:
Diagnostic Accuracy | 72 hours post-operative
  The secondary objective of the study is to estimate sensitivity (true positive rate) and specificity (true negative rate); false positive rate and false negative rate; positive predict rate, and negative predict rate using a 5-ALA dose of 20 mg/kg to delineate tumor that may provide discrimination between normal and malignant tissue intra-operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Quinones, MD, Principal Investigator — Johns Hopkins School of Medicine
Locations (2):
- United States (2):
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland